Official Title: The Health Benefits of Indoor Air Filtration Among

Children

NCT Number: NCT04835337

**Document Date: 2021-03-31** 

## **Informed Consent Form**

Dear students and parents,

We are investigators from the China Center for Disease Control and Prevention. To understand the acute impact of air pollution on children's health in China and evaluate the protective effect of air purifiers, we will conduct a randomized crossover control trial on schoolchildren. The trial consists of six visits with an interval of more than 30 days in-between. Each visit includes indoor and outdoor air pollution exposure monitoring, questionnaire surveys, physical examinations, and biological sample collection. Among them, the health examination includes growth and development indicators such as height, weight, waist circumference, and hip circumference, as well as cardiovascular and pulmonary function indicators such as blood pressure, pulse wave, electrocardiogram, lung function, exhaled nitric oxide, and exhaled carbon monoxide. The biological samples collected for each survey include: 6ml of blood, 70ml of urine, 1.5ml of saliva, 1ml of exhaled breath condensate, 1ml of oral cells, as well as feces, oral swabs, nasal swabs, skin swabs, and nails. The collected samples will be used for the detection of biomarkers, gene level methylation, and exons related to the cardiovascular, metabolic, and nervous systems. During this process, there will be no health risks or discomfort. On this basis, we provide you with feedback reports on the physical examination results of the tested children, air pollution exposure monitoring reports, personalized protective suggestions, and thank you for participating in the small gift. Based on the information you provided, we will analyze and explore changes in children's health indicators related to air pollution, and analyze their impact mechanisms to provide a basis for effective prevention and control of air pollution.

All information and test samples provided by you will be strictly confidential and will only be used for this project. We guarantee that any information you provide will not be leaked to anyone. Your name, address, and other personal information are not displayed in the database. We only record your information in code form. Your

relevant samples and data information shall be subject to confidentiality management in accordance with relevant national confidentiality regulations.

Your participation is voluntary, and if you do not agree to participate in this survey or withdraw at any time after the start, your rights will not be affected in any way; If you agree to participate in this survey and evaluation, please sign the consent statement below and leave your contact information. If you have any unclear questions during this survey, you can contact the staff:

Wang Yanwen, phone number 18811461680

Date:\_\_\_\_\_

Your cooperation is crucial for us to obtain accurate scientific data. Thank you!

| I have read and understood the above informed consent content, and I agree to participate in this survey. | |
|---|---|
| Subject signature: | |
| Date: | |
| Signature of guardian: | Phone number: |
| Date: | |
| Signature of investigator: | <u></u> |